CLINICAL TRIAL: NCT00204646
Title: Phase II Study of Neoadjuvant Dose-Intensive Chemotherapy With Adriamycin and Ifosfamide Followed by High-Dose ICE in Locally Advanced Soft Tissue Sarcomas
Brief Title: Neoadjuvant Adriamycin and Ifosfamide Plus High-Dose ICE in Patients With Soft Tissue Sarcoma (STS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: jth_005
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2007-04-20 (Estimated); Status verified 2007-04

CONDITIONS: Sarcoma, Soft Tissue
MeSH Terms: conditions — Sarcoma | interventions — Doxorubicin; Ifosfamide; Etoposide; Carboplatin

INTERVENTIONS:
Drug: Adriamycin
Drug: Ifosfamide
Drug: Etoposide
Drug: Carboplatin

SUMMARY:
Complete resection is still the only curative treatment option in patients with soft tissue sarcoma (STS). Patients with a non-resectable STS have a dismal prognosis even without evidence of metastatic disease. The aim of this trial is to determine whether neoadjuvant dose-intensive chemo-radiotherapy is a feasible and effective approach in patients with non-resectable STS.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed STS with locally advanced non-resectable disease
* Metastatic disease is allowed in case of solitary resectable metastases
* Grading according to Coindre > II°
* Measurable tumor lesions
* Age > 18 through 65 years
* Karnofsky status > 70 %
* Written informed consent

Exclusion Criteria:

* Prior chemotherapy
* Intercurrent disease interfering with the adequate administration of study medication including severe psychological disease
* Insufficient liver-, renal or bone marrow function
* Evidence of pregnancy
* Treatment within another clinical trial
* Uncontrolled viral Infections (HIV,HBV, HCV)
* other malignancies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-02; Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joerg T. Hartmann, MD, Principal Investigator — South West German Cancer Center, Medical Center II, University of Tuebingen
Locations (1):
- Medical Center II, University of Tuebingen, Tübingen, Germany